CLINICAL TRIAL: NCT05407740
Title: "ASsociation of Proteinuria and Progression of KidneY DysfunctioN in Sickle Cell Disease"
Brief Title: "Association of Proteinuria and Progression of Kidney Dysfunction in Sickle Cell Disease"Disease
Acronym: CSEG101A0FR01
Status: Completed | Type: Observational
Sponsor: Soutien aux Actions contre les Maladies du Globule Rouge (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CSEG101A0FR01
Record Dates: First submitted 2022-04-04; First posted 2022-06-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Change in Albumin to Creatinine Ratio and Glomerular Filtration Rate; Progression of Kidney Failure and or All-cause Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention study — no intervention study

SUMMARY:
To describe change in ACR and eGFR during study follow-up, and assesss the association of baseline and change in ACR and eGFR, with progression of kidney failure and/or all-cause mortality.

DETAILED DESCRIPTION:
This is a retrospective, non-interventional, secondary use of the data coming from the single-center secondary GEN-MOD study cohort at the Henri Mondor Hospital (Creteil, France). The GEN-MOD cohort includes 355 SCD patients.

The GEN-MOD data are accessible through the center's clinical and laboratory database and will be extracted and analyzed for the purpose of this study.

The enrolment in the GEN-MOD cohort lasted from 01 December 2002 until 01 March 2014. Follow-up occurred every six months and ranged from five to seventeen years and ended on 31 December 2019. The index date (baseline) for this study is the time of inclusion of patients in GEN-MOD cohort study

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years old.
* Confirmed diagnosis of SCD by Hb electrophoresis or high performance liquid chromatography. SCD genotypes HbSS, HbSβ0-thal.
* Availability of ACR and eGFR baseline records.

Exclusion Criteria:

* Patients enrolled in a chronic transfusion program.
* Patients receiving hydroxyurea treatment at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, non-interventional, secondary use of the data coming from the single-center secondary GEN-MOD study cohort at the Henri Mondor Hospital (Creteil, France). The GEN-MOD cohort includes 355 SCD patients.
  The GEN-MOD data are accessible through the center's clinical and laboratory database and will be extracted and analyzed for the purpose of this study.
  The enrolment in the GEN-MOD cohort lasted from 01 December 2002 until 01 March 2014. Follow-up occurred every six months and ranged from five to seventeen years and ended on 31 December 2019. The index date (baseline) for this study is the time of inclusion of patients in GEN-MOD cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in albumin to creatinine(ACR) and glomerular filtration rate(eGFR) | 10 years
  To describe change in ACR and eGFR during study follow-up, and assesss the association of baseline and change in ACR and eGFR, with progression of kidney failure and/or all-cause mortality

SECONDARY OUTCOMES:
Progression of kidney dysfunction | 10 years
  •To assess the association of baseline and change in ACR, and CKD progression category
Change in ACR | 10 years
  To assess potential risk factors (at baseline) for ACR elevation during study follow-up

OTHER OUTCOMES:
GFR decline | 10 years
  To assess potential risk factors (at baseline) for eGFR decline during study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: PABLO BARTOLUCCI, PROFESSOR, Principal Investigator — Soutien aux Actions contre les Maladies du Globule Rouge
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided